CLINICAL TRIAL: NCT04656795
Title: A Single Dose, Non-Randomized, Open-Label, Parallel Group Study to Investigate the Effect of Renal Impairment on the Pharmacokinetics, Safety and Tolerability of MT-7117 in Subjects With Renal Impairment Compared to Subjects With Normal Renal Function
Brief Title: PK Study in Subjects With Renal Impairment (Severe and if Required Mild & Moderate) Compared to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MT-7117-Z-101; 2020-003333-38 (EudraCT Number)
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Renal Impairment; Normal Renal Function
Keywords: PK Study in subjects with renal impairment (severe and if required mild & moderate) vs. subjects with normal renal function
MeSH Terms: conditions — Renal Insufficiency; Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Subjects with severe renal impairment (Experimental)
  Interventions: Drug: MT-7117
- Subjects with normal renal function (Experimental)
  Interventions: Drug: MT-7117
- Subjects with moderate renal impairment (Experimental)
  Interventions: Drug: MT-7117
- Subjects with mild renal impairment (Experimental)
  Interventions: Drug: MT-7117

INTERVENTIONS:
Drug: MT-7117 — MT-7117
  Other Names: dersimelagon

SUMMARY:
This is an open-label, non randomised, single-dose, study in male and female subjects with renal impairment (severe and if required mild & moderate) compared to male and female subjects with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for enrolment in the study if ALL of the following criteria apply:

For Groups 1, 2, 3 and 4

1. Subject is able to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form (ICF) and after having the opportunity to discuss the study with the Investigator or designee.
2. Male or female subjects, ≥ 18 to 80 years of age (inclusive), at the time of signing the ICF.
3. In the Investigator's opinion, subject is able to understand the nature of the study and all risks involved with participation in the study and willing to cooperate and comply with all Protocol restrictions and requirements.
4. Subjects must weigh at least 50 kg (110 pounds) and have a body mass index 18 to 35 kg/m2 both inclusive at Screening and on Day -1.
5. The subject's vital signs must be within the reference range for their age at Screening and on Day 1. Subjects must have rested for at least 5 minutes in a supine position prior to collecting blood pressure and pulse. In subjects with normal renal function, normal blood pressure is considered in the range of 90 to 145 mmHg for systolic blood pressure (SBP) and 50 to 95 mmHg for diastolic blood pressure (DBP). In subjects with renal impairment, normal blood pressure is considered in the range of 90 to 179 mmHg for SBP and 50 to 105 mmHg for DBP. Pulse rate should be between 50 to 100 beats per minutes.
6. Female subjects must not be lactating and must have a negative serum pregnancy test at Screening and on Day 1.
7. Female subjects of child bearing potential and male subjects with a partner of child bearing potential must agree to use 2 effective methods of contraception (in female subjects, one method must be highly effective.

For Group 1 (Subjects with Normal Renal Function)

1. Subjects must have an absolute eGFR of ≥ 90 mL/min, as determined by the MDRD equation, multiplied by the individual BSA according to the DuBois & DuBois equation and divided by 1.73 m2 at Screening and confirmed at Day 1 (admission to the study centre).
2. Subjects must be in good health and free from clinically significant illness or disease in the opinion of the Investigator based upon the results of medical history, physical examination, clinical laboratory tests (biochemistry, haematology, coagulation and urinalysis), vital signs and a 12 lead electrocardiogram (ECG) at Screening and Day -1.
3. Subjects with normal renal function (Group 1) will be matched in pairs by race, age (± 10 years of subject in Group 4), weight (± 10 kg of the subject in Group 4), gender and smoking status to subjects with severe renal impairment (Group 4).

For Groups 2 to 4 (Subjects with Renal Impairment)

1. Subjects must have stable renal impairment based on medical history, physical examination and clinical laboratory results. Stable renal impairment is defined as no clinically significant change in an eGFR within 3 months or longer prior to study Screening, as determined by the Investigator.
2. Subjects with renal impairment must have the following absolute eGFR values as determined by the MDRD equation, multiplied by the individual BSA according to the DuBois & DuBois equation and divided by 1.73 m2 at Screening and confirmed at Day 1 (admission to the study centre) Group 2: Mild renal impairment must have an absolute eGFR of ≥ 60 to < 90 mL/min Group 3: Moderate renal impairment must have an absolute eGFR of ≥ 30 to < 60 mL/min Group 4: Severe renal impairment must have an absolute eGFR of < 30 mL/min; not on dialysis
3. Subjects must have acceptable clinical conditions in the opinion of the Investigator based upon the results of medical history, physical examination, clinical laboratory tests (biochemistry, haematology, coagulation and urinalysis), vital signs and a 12 lead ECG at Screening and Day -1.
4. The age of subjects in Groups 2 and 3 must not be more than 10 years younger than the youngest subject in Group 1 or more than 10 years older than the oldest subject in Group 1. The weight of subjects in Groups 2 and 3 must not be more than 20% lighter than the lightest subject in Group 1 or more than 20% heavier than the heaviest subject in Group 1.
5. Subjects with mild renal impairment (Group 2) and moderate renal impairment (Group 3) will be matched by race, age, weight and gender to subjects in Group 1 (age and weight are to be matched as per inclusion criterion 4 above. It is not necessary to match subjects between Groups 2 and 3 and Group 1 in pairs, but there must be the same number of each gender and each race in each of Groups 2 and 3 as there are in Group 1).

Exclusion Criteria:

* A subject will NOT be eligible for this study if ANY of the following criteria apply:

For Groups 1, 2, 3 and 4

1. Subjects who have a known clinically significant hypersensitivity to MT-7117 or related compounds (or relevant excipients). Subjects who have a history of clinically significant hypersensitivity, intolerance, allergy or anaphylaxis to any drug compound, food or other substance unless approved by the Investigator and the Sponsor.
2. Subjects who are currently on dialysis.
3. Subjects who have any active malignancy (including melanoma but excluding basal cell carcinoma) or history of significant malignancy (including melanoma).
4. Subjects who have previously participated in a study involving MT-7117 within 6 months prior to the first dose of Investigational Medicinal Product (IMP) and/or subjects who have previously taken any other investigational drug within 2 months or 5 half-lives prior to the first dose of IMP, whichever is longer.
5. A history or presence of clinically significant neurological, haematological, psychiatric, gastrointestinal (including cholecystectomy), pulmonary or hepatic disease or other condition (with the exception of renal insufficiency for Groups 2 to 4) known to interfere with the absorption, distribution, metabolism or excretion of drugs or any condition which could place the subjects at increased risk as determined by the Investigator.
6. Clinically significant 12-lead ECG abnormalities, including subjects with corrected QT interval using Fridericia's formula (QTcF) of > 450 ms (male) and > 470 ms (female), at Screening or Day -1, confirmed by repeat assessment.
7. Subject takes non-permitted concomitant medication within 28 days (or 5 half lives of the drug, whichever is longer) of dosing on Day 1. Subjects with normal renal function are restricted from use of any concomitant medications unless discussed and agreed with the Sponsor. For renal impaired subjects, prescribed medication or over the counter (OTC) medication for treating underlying disease states or chronic medical conditions or disorders related to renal impairment are permitted as described in the protocol. If subjects with renal impairment are on any medication not listed in the protocol, this must be discussed with the Sponsor on a case-by-case basis, prior to the subject's inclusion in the study.
8. Subjects who have a positive drug screen at Screening or Day 1 (admission to the study centre), unless the positive drug screen is due to prescription drug use that is approved by the Investigator and the Sponsor.
9. Subjects who have a positive human immunodeficiency virus (HIV) antibody at Screening. Consent and counselling for this procedure will be performed according to the site's Standard Operating Procedures.
10. Subjects who have a positive test for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C antibody (HCVAb) at Screening.
11. Acute illness or infection, minor surgical procedures or trauma from within 2 weeks before Screening until administration of study drug.
12. Subjects who have a history of kidney, other organ or bone marrow transplant.
13. Subjects who have a history of major surgery within 3 months before Day 1.
14. Subjects who have a history of long QT syndrome or cardiac brady-tachy-arrhythmia.
15. Donation of 1 or more units of blood (≥ 450 mL) in the 3 months prior to Screening or plasma in the 7 days prior to Screening or platelets in the 6 weeks prior to Screening or intention to donate blood within 3 months after the final follow-up assessment.
16. Subjects who have consumed liquorice, grapefruit or grapefruit juice, orange or their associated products, within 7 days prior to study treatment on Day 1.
17. Subjects who are smokers or use tobacco or nicotine containing products (snuff, chewing tobacco, cigarettes, cigars, pipes, e-cigarettes or nicotine replacement products) and currently smoke more than 10 cigarettes or equivalent per day or are unable or unwilling to stop from 4 hours pre-dose until 6 hours post dose.
18. Subjects who are not willing to abstain from consumption of caffeine and methylxanthine (e.g., coffee, tea, cola, energy drinks or chocolates) in the 36 hours before Day 1 until completion of the post-treatment assessments on Day 4 and in the 36 hours before the Follow-up/EoS Visit on Day 8.
19. Subjects who regularly, or on average, drink more than 21 units (168 g) for males or 14 units (112 g) for females, of alcohol per week (1 unit is equivalent to 8g of alcohol).
20. Subjects with any other condition or reason that, in the opinion of the Investigator or Sponsor, would make the subject unsuitable for enrolment.
21. Subjects who test positive for Coronavirus Disease 2019 at Screening or Day -1.
22. Subject with the presence of a skin lesion suspicious for dysplastic naevus or a history of histologically proven dysplastic naevus.

Group 1 (Subjects with Normal Renal Function):

(1) Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma-glutamyl transpeptidase (GGT) or total bilirubin level (TBL) > 1.5 times upper limit of normal (ULN) during Screening or at Day 1.

For Groups 2, 3 and 4 (Subjects with Renal Impairment)

1. Use of concurrent medications, which affect the eGFR such as cephalosporin antibiotics, ascorbic acid, trimethoprim, cimetidine or quinine for at least 28 days prior to Day 1 (or 5 half-lives of the drug, whichever is longer).
2. Subject who has renal disease secondary to malignancy.
3. Subjects with acute renal failure.
4. Subject with any of the liver function test (AST, ALT, ALP and TBL) out of the following range (TBL > 1.5 × ULN, ALT and AST > 2 × ULN and ALP > 3 × ULN) at Screening or Day -1.
5. Subjects have serum albumin < 30 g/L and haemoglobin < 8 g/dL
6. Subject has not been on a stable dose of concomitant medications for the previous 28 days and/or has started new medications to treat concurrent chronic conditions in the previous 28 days (or 5 half lives of the drug, whichever is longer) prior to IMP dosing. Minor dose adjustments to the subject's regular medication may be allowed up to 14 days prior to IMP dosing after consultation with the Sponsor. This medication regimen should not change whilst the subject is enrolled in the study.
7. Any clinically significant abnormalities, other than those associated with the subject's degree of renal impairment, in biochemistry, haematology, coagulation and urinalysis results as judged by the Investigator and the Sponsor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-04 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of MT-7117 | Day 1 to 4
Area under the plasma concentration time curve from time zero to the last quantifiable concentration (AUC0-last) of MT-7117 | Day 1 to 4
Area under the plasma concentration time curve from time zero to infinity (AUC0-∞) of MT-7117 | Day 1 to 4

SECONDARY OUTCOMES:
Safety and tolerability as measured by incidence of Treatment emergent adverse events | Day -1 to Day 8
Time to maximum plasma concentration (tmax) of MT-7117 | Day 1 to 4
Apparent elimination half-time of MT-7117 in plasma (t1/2) | Day 1 to 4
Apparent oral clearance (CL/F) of MT-7117in plasma | Day 1 to 4
Apparent volume of distribution during the terminal phase (Vz/F) of MT-7117in plasma | Day 1 to 4
Unbound fraction (fu) of MT-7117 in plasma | Day 1 to 4
Maximum observed unbound plasma concentration (Cmax,u) of MT-7117 of MT-7117 | Day 1 to 4
Area under the unbound plasma concentration time curve from time zero to the last quantifiable concentration (AUC0-last, u) of MT-7117 | Day 1 to 4
Area under the unbound plasma concentration time curve from time zero to infinity (AUC0-∞, u)of MT-7117 | Day 1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (1):
- Clinical Research Services (CRS) Kiel GmbH, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ogasawara A, Ide R, Inoue S, Teng R, Kawaguchi A. Effect of Hepatic and Renal Impairment on the Pharmacokinetics of Dersimelagon (MT-7117), an Oral Melanocortin-1 Receptor Agonist. Clin Pharmacol Drug Dev. 2024 Jul;13(7):729-738. doi: 10.1002/cpdd.1413. Epub 2024 May 15. PMID 38746989